CLINICAL TRIAL: NCT02198404
Title: Pilot Study of Sedation With Propofol in Refractory Pains Due to Care in Palliative Care Unit
Acronym: PROPOPAL1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-PP-01
Record Dates: First submitted 2014-03-14; First posted 2014-07-23 (Estimated); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Refractory Pains; End of Life Patients
MeSH Terms: conditions — Pain, Intractable | interventions — Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- sedation with propofol (Experimental): propofol injection: induction with propofol at 20 mg/kg/h. When patient is sleeping, the dosage is deceased to 6 mg/kg/h
  Interventions: Drug: sedation with propofol

INTERVENTIONS:
Drug: sedation with propofol — induction with propofol at 20mg/kg/h. Then, when the patient is sleeping, dosage is decreased to 6 mg/kg/h

SUMMARY:
In the palliative care unit, certain patients suffer from pain associated with medical procedures/care which is poorly controlled by antalgics. These situations may necessitate temporary sedation to improve comfort and facilitate treatment. No proven consensus exists, either in the literature or in clinical studies conducted, on the choice of sedative agent however Midazolam is the general recommendation.

The investigators believe that Propofol could be used in this instance

DETAILED DESCRIPTION:
In the palliative care unit, certain patients suffer from pain associated with medical procedures/care which is poorly controlled by antalgics. These situations may necessitate temporary sedation to improve comfort and facilitate treatment. No proven consensus exists, either in the literature or in clinical studies conducted, on the choice of sedative agent however Midazolam is the general recommendation.

The investigators believe that Propofol could be used in this instance. The arguments in favour of Propofol include its pharmaco-kinetic characteristics and the fact that it is currently used in other circumstances. Propofol has an action delay which is more rapid that Midazolam therefore its effect is seen 1 minute after a bolus and 5 minutes after for Midazolam. The effect after a short administration lasts only a few minutes however the effect of Midazolam is more prolonged (sometimes several hours). As with Midazolam, a titrated use in weaker doses, should allow sufficient sedation, in the context which interests us, without marked secondary effects.

It is not unreasonable to think that the short action duration of Propofol could minimise respiratory risks in the hours after the treatment compared to Midazolam. With Propofol, the patient wakes as soon as the painful medical procedure has finished, with Midazolam sedation may be prolonged to several hours leading to a risk respiratory depression or secretion retention.

For these reasons; the investigators would like to verify that the use of Propofol is feasible in the context of refractory pain associated with medical procedures (dressing changes, movement during personal care tasks e.g. washing) in the palliative care unit. This is a preliminary study prior to completion of a more extensive multi-centre research project on the role Propofol could play in this situation.

ELIGIBILITY:
Inclusion Criteria:

* patients hospitalized in palliative care unit
* dying terminally patients
* pains resisting to fentanyl and MEOPA (Melange equimolaire Oxygène protocyde d'Azote) (EMONO = equimolar mixture of oxygene and nitrous oxide)

Exclusion Criteria:

* contra-indication to soya
* contra-indication to egg lecithin
* Respiratory insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-06-20; Primary Completion 2015-09-29 (Actual); Study Completion 2015-09-29 (Actual)

PRIMARY OUTCOMES:
Feasability of the care without largely pain | at inclusion (day=0), after the care
  The nurse assess if the care could be done without largely pain for the patient. The answer would be "yes" or "not"

SECONDARY OUTCOMES:
asleep delay | at the inclusion (day=0), delay between sleep-inducing medicine injection and asleep
  time in minutes between injection of propofol and sleep of patient

CONTACTS AND LOCATIONS:
Overall Officials: CIAIS Jean-François, PhD, Principal Investigator — Nice University Hospital
Locations (1):
- Nice University Hospital, Nice, France